CLINICAL TRIAL: NCT05674591
Title: Cognitive Processing Therapy for the Treatment of Depression, Anxiety, PTSD, and Difficulties in Emotion Regulation in Syrian Females Exposed to Intimate Partner Violence
Brief Title: Cognitive Processing Therapy in Syrian Women Exposed to IPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-2021
Record Dates: First submitted 2022-12-14; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anxiety; PTSD
Keywords: Cognitive Processing Therapy; Syrian women; Mental health
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: The current study is a clinical trial, including the repeated assessments of a single sample of Syrian women. Pre-treatment, posttreatment and 12-month posttreatment assessments were conducted on participants. PTSD severity, depression, anxiety and difficulties in emotion regulation will be assessed as outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive Processing Therapy (Experimental): Cognitive Processing Therapy (CPT) is a manual-guided therapy that incorporates cognitive processing techniques to relieve PTSD symptoms (Resick et al., 2016). Each group session will be 90 to 120 minutes long and will be occur once each week for 12 weeks.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — The CPT therapist will teach the patient about PTSD, depression, and anxiety, and outline the treatment regimen and rationale for its effectiveness. In the initial sessions, women will be asked to express their impact statements on the intimate partner violence to which they had been subjected. Women will be taught how to differentiate between events, thoughts, and emotions, as well as their interrelationships. Thoughts of self-blame and other misconceptions of the situation will be addressed using Socratic questioning. Women will be instructed on how to detect and counteract negative thoughts, as well as how to communicate more effectively. Women will be encouraged to evaluate negative thinking relating to five themes: safety, trust, power/control, self-esteem, and intimacy. During the final sessions, their impact statements on the violence to which they had been subjected will be altered to include emotional and cognitive insights obtained during the CPT.
  Other Names: CPT

SUMMARY:
This study aims to explore the efficacy of cognitive processing therapy (CPT) in treating depression, anxiety, PTSD, and difficulties with emotion regulation in Syrian females who have suffered intimate partner violence (IPV). Clinicians will conduct interviews with women and request that they complete the CAPS, Beck Depression Inventory II, Beck Anxiety Inventory, and DERS during pretreatment, posttreatment, and at the 12-month follow-up

DETAILED DESCRIPTION:
This study aims to explore the efficacy of cognitive processing therapy (CPT) in treating depression, anxiety, PTSD, and difficulties with emotion regulation in Syrian females who have suffered intimate partner violence (IPV). Clinicians will conduct interviews with women and request that they complete the CAPS, Beck Depression Inventory II, Beck Anxiety Inventory, and DERS during pretreatment, posttreatment, and at the 12-month follow-up. Cognitive processing therapy (CPT) may have a substantial therapeutic benefit in the treatment of depression, anxiety, PTSD, and difficulties in emotion regulation among Syrian females who have suffered intimate partner violence.

ELIGIBILITY:
Inclusion Criteria:

* being a Syrian female who currently exposes to intimate partner violence,
* lives in Egypt
* has a good knowledge of English language because all assessments and therapy materials are in English.

Exclusion Criteria: having:

* cognitive difficulties
* schizophrenia (or any other psychotic disorders).

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 30 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Women's Health and Domestic Violence against Women questionnaire | At first interview, pretreatment
  Version 11 of the WHO Multi-Country Study on Women's Health and Domestic Violence against Women questionnaire (WHO, 2005). This instrument comprises of an informed consent form, a household questionnaire, and a 1-item questionnaire regarding the circumstances of women. The WHO Multi-country Study on Women's Health and Domestic Violence assesses whether women have been subjected to any kind of intimate partner violence throughout their lives. The four components of intimate partner violence are physical, sexual, emotional, and controlling violence. Indicators were dichotomous, with 1 indicating whether or not the individual was a victim of IPV (1 = "Yes", 0 = "No"). Women were asked a number of questions on whether they had ever encountered a variety of behaviours belonging to one of the four groups. For each act of violence, participants will be required to identify whether it had occurred in their lives and how frequently it had occurred
Change from Baseline on Clinician-Administered PTSD Scale at 3 months and at 12 months | baseline (pre-intervention), posttreatment (immediately after the intervention, an average of 3 months), 12-months after the intervention
  Currently, the CAPS-5 (Weathers et al., 2015) is the global standard for PTSD evaluation and is used to evaluate PTSD symptoms. This 30-item structured interview was created by the National Centre for PTSD of the US Department of Veterans Affairs. Generally, the interview may be conducted in 45 to 60 minutes. Each CAPS-5 question addresses both the frequency and severity of each PTSD symptom. These questions have been categorized. Each criteria comprises many questions, and at the end, the points for each criterion are totaled together. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms. The cutoff score for CAPS-5 is 45. Higher scores on CAPS mean a worse outcome. Improvement was defined as a 5 point reduction in the overall CAPS-5 scores. Remission was defined as loss of diagnosis and no longer having any PTSD symptoms according to minimum severity scores on CAPS-5 (< 12)
Change from Baseline on Beck Depression Inventory II scores at 3 months and at 12 months | baseline (pre-intervention), posttreatment (immediately after the intervention, an average of 3 months), 12-months after the intervention
  BDI-II measured depression symptoms. BDI-II is a 21-item self-report assessment measuring depressive attitudes and symptoms (Beck et al., 1996). BDI-II takes 10 minutes. Minimal range=0-13, mild depression=14-19, moderate depression=20-28, and severe depression=29-63. BDI-II is reliable and valid (Beck et al., 1996)
Change from Baseline on Beck Anxiety Inventory scores at 3 months and at 12 months | baseline (pre-intervention), posttreatment (immediately after the intervention, an average of 3 months), 12-months after the intervention
  BAI measures somatic anxiety symptoms as anxiousness, dizziness, and inability to relax (Beck et al., 1988). It takes 10 to 15 minutes to finish 21 items. Four-point Likert scale answers vary from zero to three (severely). The total score for all 21 symptoms ranges from 0 to 63 points.
  A score of 0-7 indicates "little" anxiety, 8-15 "mild," 16-25 "moderate," and 26-63 "severe" (Beck & Steer 1990)
Change from Baseline on Difficulties Emotion Regulation scale scores at 3 months and at 12 months | baseline (pre-intervention), posttreatment (immediately after the intervention, an average of 3 months), 12-months after the intervention
  The DERS was created by Gratz and Roemer (2004) and consists of a 36-item self-report questionnaire that evaluates the difficulty in regulating emotions. Bjureberg et al. (2016) created a 16-item abbreviated version of the DERS later on. There are three items about nonacceptance, three items regarding difficulties participating in goal-directed actions, three things regarding impulsivity, five items regarding trouble utilizing emotion regulation strategies, and two items regarding emotional clarity Items are rated on a scale of 1 ("almost never [0-10%]") to 5 ("almost always [91-100%]"). Higher scores indicate more difficulty in emotion regulation. Higher scores on DERS mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amani Elbarazi, PhD, Principal Investigator — The British University in Egypt
Locations (1):
- The British university in Egypt, Cairo, Egypt